CLINICAL TRIAL: NCT05954247
Title: Bioequivalence Study for the Safety and the Pharmacokinetics of DWJ1543 in Healthy Adult Volunteers Under Fasting Conditions
Brief Title: Bioequivalence Study for the Safety and the Pharmacokinetics of DWJ1543 in Healthy Adult Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DW_DWJ1543101
Record Dates: First submitted 2023-07-12; First posted 2023-07-20 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: DWJ1543 (Experimental)
  Interventions: Drug: DWJ1543
- Intervention: DWC202216 (Experimental)
  Interventions: Drug: DWC202216

INTERVENTIONS:
Drug: DWJ1543 — DWJ1543
  Arms: Intervention: DWJ1543
Drug: DWC202216 — DWC202216
  Arms: Intervention: DWC202216

SUMMARY:
This study aims to evaluate the safety and pharmacokinetic characteristics after administration of DWJ1543 in healty adult volunteers.

DETAILED DESCRIPTION:
The study design is a Randomized, Open-label, Oral, Single-dose, Two-way crossover study. The patients were randomly assigned to each group. Primary endpoint was Cmax and AUClast of DWP16001. Secondary endpoints were AUCinf, AUClast, Tmax, t1/2, CL/F, and Vd/F of DWJ1543.

ELIGIBILITY:
Inclusion Criteria:

* Over 19 year old
* Healthy adult volunteers

Exclusion Criteria:

* Eye disorders including cataracts
* Respiratory disorders including interstitial lung disease and pneumonitis and venous thromboembolic disorders

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Maximum plasma concentration at steady-state(Cmax,ss) of DWJ1543 | At pre-dose (0 hour), and post-dose 1 to 120 hour.
Area under the curve from the time of dosing to the last measurable concentration(AUClast) of DWJ1543 | At pre-dose (0 hour), and post-dose 1 to 120 hour.